CLINICAL TRIAL: NCT04303806
Title: Effect of Rosuvastatin on Sever Preeclampsia Induced Inflammatory Response
Brief Title: Effect of Rosuvastatin on the Clinical Features of Preeclampsia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mansour, assistant lecturer on anasthesia and icu department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: rosuvastatin on preeclampsia
Record Dates: First submitted 2019-09-23; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: . They will be randomly allocated into two equal groups of 40 parturient each: Group 1: 40 preeclamptic parturient receive 20 mg rosuvastatin orally once daily.
  Group 2: 40 preeclamptic parturient receive 40 mg rosuvastatin orally once daily
Who Masked: Participant, Investigator
Masking Description: computer generated randomization will be conducted in a Women's Health Hospital, Assuit University. Neither the doctor "investigator" nor the participant "parturient" will be aware of the group allocation or the drug used. The study drugs will be prepared by one of the supervisor anesthesia (not included in the procedure, observation or in data collection)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 40 preeclamptic parturient receive 20 mg rosuvastatin orally once daily.
  Interventions: Drug: rosuvastatin
- Group 2 (Experimental): 40 preeclamptic parturient receive 40 mg rosuvastatin orally once daily.
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — receive rosuvastatin orally once daily.

SUMMARY:
The primary outcome will be the effect of rosuvastatin on the resolution of biochemical features associated with severe PE (↑CRP and IL6).

.

DETAILED DESCRIPTION:
Preeclampsia is a multisystem disorder that complicates 3-5% of pregnancies and remains a major cause of maternal, fetal, and neonatal morbidity and mortality.(1)

Preeclampsia is characterized by the development of new onset hypertension (HTN) and the establishment of proteinuria. Other signs and symptoms that accompany the disease include: headache, visual disturbances, epigastric or abdominal pain, weakness, altered mental status, HELLP syndrome (2) dyspnea and edema (American College of Obstetricians and Gynecologists and Task Force on Hypertension in Pregnancy, 2013).

Previous preeclamptic pregnancy, family history of preeclampsia, late age of maternity (>40 years), multiple gestation, obesity, diabetes mellitus and history of thrombophilia have been identified as predisposing risk factors (American College of Obstetricians and Gynecologists and Task Force on Hypertension in Pregnancy, 2013). In particular, the presence of HTN and chronic renal impairment before gestation has been strongly correlated to the development of preeclampsia later during pregnancy (Foo et al., 2015).

Preeclampsia can result in a great number of severe and, in some cases, fatal short- and long-term consequences affecting both the mother and the fetus. Maternal complications include cardiometabolic disorders (diabetes, ischemic heart disease, metabolic syndrome), cerebrovascular disease (stroke, intracranial bleeding), neurologic abnormalities (eclamptic seizures) and renal impairment (Ramsay et al., 2003; Wilson et al., 2003; Haukkamaa et al., 2004; Funai et al., 2005).

Fetal outcomes include intrauterine growth restriction (IUGR), prematurity and higher risk of developing HTN, obesity, metabolic syndrome, dyslipidemias, and cardiovascular disease (Lo et al., 2013; Nice guidelines, 2016).

There is evidence from several studies that preeclampsia is accompanied by endothelial injury. This injury results in abnormal vascular relaxation and platelet activation and is associated with inflammation and oxidative imbalance. (5) The activation of the inflammatory cascade that occurs in normal pregnancy is further exaggerated in preeclampsia. Markers of inflammation, such as high-sensitivity C-reactive protein (hs-CRP), are elevated in patients who later develop preeclampsia. In addition, preeclampsia is associated with elevated cytokines such as tumor necrosis factor-α, interleukin-6 (IL-6), and IL-12. These activate the inflammatory cascade and increase free radical generation and oxidative stress, thus contributing to endothelial injury. (6)

Delivery of the fetus is the only efficient therapy (Everett et al., 2012; Gangooly et al., 2014; Nice guidelines, 2016(10. Nice guidelines (2016). Hypertension in Pregnancy: Diagnosis and Management |

1-Guidance | Guidance and guidelines | NICE. [cited 2016 May 27]. Available at: https://www.nice.org.uk/guidance/cg107/chapter/1-guidance ) ). If the gestational age is less than 34 weeks and the BP can be sufficiently controlled with the absence of other symptoms, pregnancy can be prolonged in order to avoid prematurity complications for the fetus. The main therapeutic goal in preeclampsia is the management of HTN, aiming for SBP of 140-150 mmHg and DBP of 80-100 mmHg (Nice guidelines, 2016 10. Nice guidelines (2016). Hypertension in Pregnancy: Diagnosis and Management |

1-Guidance | Guidance and guidelines | NICE. [cited 2016 May 27]. Available at: https://www.nice.org.uk/guidance/cg107/chapter/1-guidance). Oral antihypertensive therapy including a-methyldopa, calcium channel blockers, b-blockers and labetalol, coupled with antiplatelet agents and magnesium sulfate are considered as a therapy in hypertensive disorders in order to limit maternal and fetal complications (Sandrim et al., 2008; Nice guidelines, 2016 12. Sandrim, V. C., Palei, A. C., Metzger, I. F., Gomes, V. A., Cavalli, R. C., and Tanus-Santos, J. E. (2008). Nitric oxide formation is inversely related to serum levels of antiangiogenic factors soluble fms-like tyrosine kinase-1 and soluble endogline in preeclampsia. Hypertension 52, 402-407. doi: 10.1161/ HYPERTENSIONAHA.108.115006

).

Statins are 3-hydroxy-3-methylglutaryl coenzyme A (HMG CoA) reductase inhibitors that are effective in the reduction of total and LDL cholesterol.3 They prevent initial cardiovascular and subsequent cardiovascular events in ischemic heart disease patients, irrespective of the cholesterol concentration.5,6

There has been recent interest in the use of statins to treat preeclampsia. Notably, evidence has emerged that statins have vasoprotective properties independent of their effects in lowering serum cholesterol.8,9 ) Statins also correct the imbalance in the Th1/Th2 cytokine responses observed in preeclampsia (statins decrease Th1 proinflammatory cytokines, such as TNF-α, IL-1, IL-2, IFN-γ, and increase Th2 antiinflammatory cytokines such as IL-4, IL 10). (23) Cudmore et al10 showed that simvastatin significantly reduced sFlt-1 secretion from placenta and endothelial cells. Unfortunately, simvastatin may not be acceptable for use during pregnancy. It has a category X rating in light of observational studies, demonstrating an association with fetal malformations if administered during the first trimester.11,12 Some have proposed that rosuvastatin may be a more promising therapeutic candidate given its safety profile could be better than simvastatin.

Unlike simvastatin, which is hydrophobic, rouvastatin is hydrophilic, meaning it may less readily cross through the placenta to the fetus.11,13 Transplacental transfer of statins depends on their plasma concentration; their binding to plasma proteins; their molecular weight, lipophilicity and ionization state; and their capacity to bind to placental transport proteins. Pravastatin and rosuvastatin are relatively hydrophilic (which, in theory, reduces their transplacental passage) and not significantly metabolized by CYP enzymes.[20] Cohort studies have shown that administration of lipophilic statins have increased fetal malformation risk; however, hydrophilic statins, including rosuvastatin, have not been associated with an increased risk.11

Rosuvastatin is a fully synthetic HMG-CoA reductase inhibitor. It belongs to a new generation of methane-sulphonamide pyrimidine and N-methane sulfonyl pyrrole-substituted 3, 5- dihydroxy-heptenoates. Although the characteristic statin pharmacophore remains similar to other statins, the addition of a stable polar methane-sulphonamide group provides low lipophilicity and enhanced ionic interaction with HMG-CoA reductase enzyme thus improving its binding affinity to this enzyme.16-18((16. White CM. A review of the pharmacologic and pharmacokinetic aspects of rosuvastatin. J Clin Pharmacol. 2002; 42: 963-70.

18. McTaggart F. Comparative pharmacology of rosuvastatin. Atherosclerosis. 2003; 4:9-14))

As observed with other statins, rosuvastatin has pleiotropic effects independent of HMG-CoA reductase inhibition. These include improvements in endothelial function, anti-inflammatory, antithrombotic and anti-oxidant effects.27((27. Grosser N, Erdmann K, Hemmerle A, et al. Rosuvastatin upregulates the antioxidant defense protein heme oxygenase-1. Biochem Biophys Res Commun. 2004; 325: 871-6)) Statins improve endothelial function by increasing the production of endothelial nitric oxide and reducing the production of oxygen derived free radicals. Rosuvastatin reduces high sensitivity C reactive protein (hsCRP) which is a marker of inflammation and an independent cardiovascular risk predictor and other inflammatory markers.28(28. Mayer C, Gruber HJ, Landl EM, et al. Rosuvastatin reduces interleukin- 6-induced expression of C-reactive protein in human hepatocytes in a STAT3- and C/EBP-dependent fashion. Int J Clin Pharmacol Ther. 2007; 45: 319-27)) It inhibits platelet aggregation to leukocytes which inhibit formation of clots in injured endothelium.29 (29. Laumen H, Skurk T, Hauner H, et al. The HMG-CoA reductase inhibitor rosuvastatin inhibits plasminogen activator inhibitor-1 expression and secretion in human adipocytes. Atherosclerosis. 2008;196: 565-73)

Approximately 90% of rosuvastatin is protein bound mainly to albumin. It is less lipophilic than other statins and has a plasma half life of 19 hours which is longer than atorvastatin (15 hours) and simvastatin (2-3 hours). It is primarily eliminated in the faeces (90%) compared with 10% renal excretion. Approximately 72% of absorbed rosuvastatin is eliminated in bile and 28% via renal excretion.33(33. Martin PD, Warwick MJ, Dane AL, et al. Metabolism, excretion, and pharmacokinetics of rosuvastatin in healthy adult male volunteers. Clin Ther. 2003;25:2822-35.) As the circulating half life is 19 hrs it can be taken once daily at any time of the day regardless of meals.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35 years.
* Singleton nonanomalous pregnancy (confirmed with an ultrasound examination).
* Normal lipid profile and normal liver transaminases.
* WBCs (4-11*103/mm3).
* CRP < 3 mg/L.

Exclusion Criteria:

* Parturient's refusal.
* Women with history of cardiac, respiratory, renal, neurologic or endocrine diseases.
* Contraindications for statin therapy (eg, hypersensitivity to rosuvastatin, recent or active liver disease).
* Concomitant therapy with fibrates, niacin, cyclosporine, clarithromycin, or erythromycin.
* Inability to tolerate oral medications secondary to severe nausea and vomiting of pregnancy.
* Multifetal gestation or fetal demise.
* Fetal abnormalities.
* Emergency surgeries.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the effect of rosuvastatin on the clinical features of preeclampsia | baseline
  The primary outcome will be the effect of rosuvastatin on the resolution of biochemical features associated with severe PE (↑CRP and IL6).

IPD SHARING:
Plan to Share IPD: Yes